CLINICAL TRIAL: NCT05276284
Title: TEMPLE - Thiopurine Enhanced Mutations for PD-1/Ligand-1 Efficacy
Brief Title: Thiopurine Enhanced Mutations for PD-1/Ligand-1 Efficacy
Acronym: TEMPLE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kristoffer Rohrberg (Other)
Responsible Party: Sponsor-Investigator, Kristoffer Rohrberg, Sponsor- investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEMPLE01
Record Dates: First submitted 2022-02-04; First posted 2022-03-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — atezolizumab; Mercaptopurine; Thioguanine

STUDY DESIGN:
Intervention Model Description: The TEMPLE study is a single-center prospective phase Ib and II trial to determine the safety, tolerability and efficacy of Atezolizumab given in combination with thiopurine therapy in patients with advanced and/or metastatic solid tumors with an intermediate tumor mutational burden.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEMPLE (Experimental): Study drugs: Atezolizumab, 6-mercaptopurine and 6-thioguanine
  Interventions: Combination Product: Atezolizumab, 6-mercaptopurine, 6-thioguanine

INTERVENTIONS:
Combination Product: Atezolizumab, 6-mercaptopurine, 6-thioguanine — Combination therapy with Atezolizumab, 6-mercaptopurine and 6-thioguanine

SUMMARY:
The TEMPLE study is a single-center prospective phase Ib and II trial to determine the safety, tolerability and efficacy of Atezolizumab given in combination with thiopurine therapy (6-mercaptopurine and 6-thioguanine) in patients with advanced and/or metastatic solid tumors with an intermediate tumor mutational burden.

Maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) will be determined in a single armed, open label phase Ib trial with a fixed dose of Atezolizumab in combination with thiopurine therapy with a dose-limiting toxicity (DLT) period of 4 weeks. A total of 27-39 patients will be enrolled in the TEMPLE study. Phase Ib will enroll 3-18 patients depending on the number of DLTs and need for dose de-escalation. Data from patients treated in the phase Ib study at RP2D will be included when assessing endpoints in the phase II part of the study. Phase II will enroll a total of 27 patients (including 3-6 patients treated at RP2D in the phase I part of the trial) in a Simon's 2 stage design (13 in stage 1 and 14 in stage 2).

DETAILED DESCRIPTION:
INTRODUCTION:

Immune checkpoint inhibitors (ICI) have revolutionized treatment of several cancer types. However, many patients fail to respond. A prerequisite for response is the presence of neoepitopes on cancer cells that trigger the immune system, and the likelihood hereof increases with the number of mutations in the cancer. The thiopurines 6-mercaptopurine (6MP) and 6-thioguanine (6TG) are prodrugs that are converted into cytotoxic metabolites that are incorporated into DNA (DNA-TG) and cause DNA-damage through futile DNA mismatch repair attempts. 6MP and 6TG have been used for more than 50 years for long-term treatment of hematological cancers. In leukemia, high levels of DNA-TG are associated with higher cure rates. A recent pilot study has shown that combination therapy with 6MP and 6TG significantly increases DNA-TG levels and that the drug combination is safe and tolerable. The higher DNA-TG levels most likely increase the mutational burden and thus presence of neoepitopes that activate cytotoxic T-cell responses.

The TEMPLE project will apply the innovative thiopurine combination strategy to increase the mutational burden, presence of neoepitopes and thus proportion of patients with incurable solid cancers that respond to treatment with ICIs.

STUDY DESIGN:

The TEMPLE study is a single-center prospective phase Ib and II trial to determine the safety, tolerability and efficacy of Atezolizumab given in combination with thiopurine therapy in patients with advanced and/or metastatic solid tumors with an intermediate tumor mutational burden. Maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) will be determined in a single armed, open label phase Ib trial with a fixed dose of Atezolizumab in combination with thiopurine therapy. In the phase Ib part of the study, patients will start treatment with investigational medicinal products:

1. 6-mercaptopurine (6MP) 50 mg/m2 orally taken once a day,
2. 6-thioguanine (6TG) 12.5 mg/m2 orally taken once a day, and
3. Atezolizumab 1200 mg every 3 weeks

The combination of thiopurines and Atezolizumab will be administered in 21-day cycles. The DLT evaluation period will be four weeks. Patients will be included in a modified 3+3 design. 3-18 patients are expected to be enrolled in the phase Ib study, depending on observed DLTs. Phase II be an open label, single arm phase II trial enrolling additional patients up to a total of 27 patients treated at RP2D in a Simon's 2 stage design (13 in stage 1 and 14 in stage 2).

All three study drugs are already approved for within hospital use in Denmark and the Summary of Product Characteristics (SmPCs) will be used in assessment of possible undesirable effects during the study. Patients will be monitored closely for adverse events using the NCI CTCAE v 5.0. If patients develop toxicity, the dose may be modified or discontinued. All dosing interruptions and modifications should be based on the worst preceding toxicity. Patients will be monitored continuously, and dose modifications or interruptions will occur based on the observed toxicity. For Atezolizumab, no dose reduction is permitted, but infusions may be omitted. Dose modifications may be implemented to manage toxicities for 6MP and 6TG.

Patients will continue treatment until progression disease, death, development of unacceptable toxicity or withdrawal of consent. Patients can be treated for a maximum of 2 years with option to re-challenge upon progression or relapse for those responding.

ELIGIBILITY:
Inclusion Criteria:

The patient MUST MEET ALL the following criteria to be enrolled in the study:

1. Signed written informed consent.
2. Age ≥ 18 years.
3. Performance status (WHO) of 0-1.
4. Histologically confirmed advanced and/or metastatic solid tumors for which standard curative measures do not exist.
5. Radiologically measurable disease according to RECIST v1.1.
6. Life expectancy estimated by the Investigator to be ≥12 weeks.
7. Metastatic Lesion(s) or primary tumour accessible for biopsy
8. Intermediate tumor mutational burden of 5-10 mutations/mb
9. Adequate organ function assessed by screening laboratory values:

   1. Absolute lymphocyte count ≥ 0.5 x 109/L
   2. Neutrophils ≥ 1.5 x 109/L
   3. Platelets ≥ 100 x 109/L. For patients with primary hepatocellular carcinoma platelet counts ≥65 x 109/L is allowed.
   4. Hemoglobin ≥ 90 g/L (5.6 mmol/L) and at least 4 weeks since blood transfusion
   5. Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or calculated by Cockroft-Gault formula or directly measured creatinine clearance ≥ 50 mL/min at screening
   6. AST ≤ 3 x ULN without, and ≤ 5 x ULN with hepatic metastasis
   7. Bilirubin ≤ 1.5 x ULN (except patients with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL)
10. Ability to take oral medications.
11. Woman of childbearing potential must have been tested negative in a serum pregnancy test within 5 days prior to study drug initiation.
12. Male and female patients who have the potential to reproduce must agree to use a highly effective method of birth control (i.e., pregnancy rate of less than 1 % per year) during the study and for 5 months after the discontinuation of study medication. Women must refrain from donating eggs and men must refrain from donating sperm during this same period.

Exclusion Criteria:

Any of the following :

1. Pregnancy, lactation, or breastfeeding.
2. History or clinical evidence of central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases, unless they have been previously treated, are asymptomatic, and have had no requirement for steroids or anticonvulsants in the last 14 days prior to Screening.
3. Deficiency in thiopurine methyltransferase (TPMT) or NUDT15.
4. Use, or have used, any concomitant anti-cancer medications within the previous 30 days or 5 half-lives of the medication (whichever is shortest) prior to first dose (bisphosphonates, denosumab and androgen deprivation therapies such as LHRH (GnRH) agonists are allowed if patient is on stable treatment for at least 4 weeks prior to first dose). Limited field radiotherapy for palliative purpose is allowed at any time.
5. Participants with immune-related adverse events attributed to prior immunomodulatory therapy must have resolved to Grade ≤ 1 (according to NCI CTCAE v 5.0) or baseline other than adverse events that are clinically non-significant and/or stable on supportive therapy, and are not expected to interfere with treatment in the study such as:

   1. Grade ≤ 2 alopecia, asthenia, dermatologic events.
   2. Grade ≤ 2 anemia if hemoglobin ≥ 90 g/L (5.6 mmol/L)
   3. Grade 2 (> 1.5-2.0 x ULN) asymptomatic amylase and/or lipase elevation with no abdominal pain and no characteristic CT findings. However, weekly monitoring of amylase and lipase is required in this case.
6. Be an organ transplant recipient.
7. Have a history of prior other malignancy (with the exception of localized prostate cancer, adequately treated basal skin cancer or carcinoma in-situ of the cervix) within 2 years prior to first dose.
8. Have a severe autoimmune disorder requiring treatment during the last 12 months prior to first dose. Diabetes on stable anti-diabetic medication, hypothyroidism and adrenocortical deficiency on stable substitution therapy are allowed.
9. Be on chronic therapy with systemic immunosuppressant medication (inhaled, intra articular and low dose systemic corticosteroids, e.g. 7.5 mg or less prednisolone per day is allowed, provided that treatment has been unchanged for at least 4 weeks prior to first dose of IMP).
10. Known HIV, active hepatitis B or hepatitis C infection.
11. Participants with a history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or known hypersensitivity to Chinese hamster ovary cell products or to any component of the Atezolizumab formulation
12. Any condition that, in the opinion of the Investigator, would place the patient at increased risk or preclude the patient's compliance with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 3-6 months
  Type and number of adverse events
Dose limiting toxicities | 28 days
  Dose limiting toxicities (DLTs) and the MTD for determination of RP2D of Atezolizumab, 6TG and 6MP
Best overall response | One year
  Complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), unconfirmed (iUPD) and confirmed PD (iCPD), assessed according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1

SECONDARY OUTCOMES:
Progression Free Survival | Two years
  Survival time without progression
Overall Survival | Two years
  Survival time of participants
Duration of response | Two years
  Time from initial time of response according to RECIST 1.1 until progression, censoring or death.

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer S Rohrberg, MD PhD, Principal Investigator — MD, Phd, Consultant, Head of Phase 1 Unit, Department of Oncology, Rigshospitalet
Locations (1):
- University Hospital of Copenhagen, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Nazerai L, Willis SC, Yankilevich P, Di Leo L, Bosisio FM, Frias A, Bertolotto C, Nersting J, Thastrup M, Buus S, Thomsen AR, Nielsen M, Rohrberg KS, Schmiegelow K, De Zio D. Thiopurine 6TG treatment increases tumor immunogenicity and response to immune checkpoint blockade. Oncoimmunology. 2022 Dec 17;12(1):2158610. doi: 10.1080/2162402X.2022.2158610. eCollection 2023. PMID 36545256